CLINICAL TRIAL: NCT05687409
Title: Alterations in the Intestinal Microbiome and Metabolic Profile of Patients With Cirrhosis Supplemented With Lactulose, Clostridium Butyricum, and Bifidobacterium Longum Infantis: a Randomized Placebo-controlled Trial
Brief Title: Synbiotics Interventions for Managing Cirrhosis and Its Complications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: wuzhongwenzju
Record Dates: First submitted 2022-11-25; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-11

CONDITIONS: Cirrhosis, Liver; Metagonimiasis
Keywords: Cirrhosis, Liver; Synbiotics
MeSH Terms: conditions — Liver Cirrhosis; Trematode Infections | interventions — entecavir; Probiotics; Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A 10-g packet of lactulose oral solution and three capsules of probiotics +entecavir group (Experimental): 10-g packet of lactulose oral solution and three capsules of probiotics +entecavir group:Adults with histologically confirmed stable cirrhosis and BMI < 25 kg m-2 were enrolled and assigned to receive boxes labeled A or B: one for the synbiotic, including a 10-g packet of lactulose oral solution and three capsules of probiotics (each containing > 4.2×106 CFU Clostridium butyricum and > 4.2×105 CFU Bifidobacterium longum infantis). Participants orally administered the contents three times daily after meals.
  Entecavir 5mg, once a day. All of the above lasted for six months.
  Interventions: Drug: Entecavir 0.5 mg; Drug: A 10-g packet of lactulose oral solution and three capsules of probiotics
- A 10-g packet of glucose oral solution and three capsules of starch+entecavir group (Placebo Comparator): A 10-g packet of glucose oral solution and three capsules of starch+entecavir group:Adults with histologically confirmed stable cirrhosis and BMI < 25 kg m-2 were enrolled and assigned to receive boxes labeled A or B: one for the synbiotic, including a 10-g packet of lactulose oral solution and three capsules of probiotics (each containing > 4.2×106 CFU Clostridium butyricum and > 4.2×105 CFU Bifidobacterium longum infantis). Participants orally administered the contents three times daily after meals.
  Entecavir 5mg, once a day. All of the above lasted for six months.
  Interventions: Drug: Entecavir 0.5 mg; Dietary Supplement: A 10-g packet of glucose oral solution and three capsules of starch

INTERVENTIONS:
Drug: Entecavir 0.5 mg — Orally administered Entecavir 0.5 mg, once a day. For six months
Drug: A 10-g packet of lactulose oral solution and three capsules of probiotics — A 10-g packet of lactulose oral solution and three capsules of probiotics (each containing > 4.2×106 CFU Clostridium butyricum and > 4.2×105 CFU Bifidobacterium longum infantis).
  Participants orally administered the contents three times daily after meals. For six months.
  Arms: A 10-g packet of lactulose oral solution and three capsules of probiotics +entecavir group
Dietary Supplement: A 10-g packet of glucose oral solution and three capsules of starch — A 10-g packet of glucose oral solution and three capsules of starch. Participants orally administered the contents three times daily after meals. For six months.
  Arms: A 10-g packet of glucose oral solution and three capsules of starch+entecavir group

SUMMARY:
Background Liver cirrhosis is commonly accompanied by intestinal dysbiosis and metabolic defects. Many clinical trials have shown microbiota-targeting strategies represent promising interventions for managing cirrhosis and its complications. However, the influences of the intestinal metagenomes and metabolic profiles of patients have not been fully elucidated.

Methods administered lactulose, Clostridium butyricum, and Bifidobacterium longum infantis as a synbiotic and used shotgun metagenomics and non-targeted metabolomics to characterize the results.

ELIGIBILITY:
Inclusion Criteria:

* ① Hepatitis B cirrhosis was diagnosed by clinical biochemistry and imaging.

  * CTP rating is a-b.

    * There was a previous liver cirrhosis complication, including ascites, spontaneous peritonitis, massive gastrointestinal bleeding, liver coma, etc.

      * Over 18 years old. ⑤ Under 90 years old.

        * The patient or family member signs the informed consent form.

Exclusion Criteria:

* ① The CTP of liver cirrhosis was evaluated as grade C.

  * Other types of cirrhosis such as primary biliary cirrhosis.

    * Pregnancy status. ④ Have a history of diabetes, renal insufficiency, gastrointestinal surgery, etc.

      * Antibiotics, PPI preparations and microecological preparations (including yogurt) have been used in the past 8 weeks.

        * Have a history of narcotic drug abuse, drug abuse, or mental illness. ⑦ Patients and their families do not agree to sign the informed consent form. ⑧ Under 18 years old or over 90 years old.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-24 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Liver CT to assess cirrhosis in 70 cirrhotic participants | Up to 11 months
  Liver CT was used to evaluate the liver cirrhosis of 70 cirrhotic participants
Assessing the intestinal microbiota of 120 cirrhotic and healthy participants through fecal metagenomics | Up to 12 months
  fecal metagenomics was used to assess the intestinal microbiota of participants.
Metabolomics to assess the metabolites of the 120 cirrhotic and healthy participants' intestinal microbiota including polyketides(Casimiroedine μmol/L),Benzenoids(Olmesartan μmol/L),Organoheterocyclic compounds(Amlexanox μmol/L) and etc. | Up to 12 months
  Metabolomics was used to assess the metabolites of the participants' intestinal microbiota.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
share date: within 6 months after project finish. Website: Resman. http://www.medresman.org.cn/pub/cn/proj/search.aspx

REFERENCES:
- [Derived] Lu H, Zhu X, Wu L, Lou X, Pan X, Liu B, Zhang H, Zhu L, Li L, Wu Z. Alterations in the intestinal microbiome and metabolic profile of patients with cirrhosis supplemented with lactulose, Clostridium butyricum, and Bifidobacterium longum infantis: a randomized placebo-controlled trial. Front Microbiol. 2023 Apr 26;14:1169811. doi: 10.3389/fmicb.2023.1169811. eCollection 2023. PMID 37180228